CLINICAL TRIAL: NCT06614504
Title: A Randomized Controlled Trial of Reduced Nicotine Cigarettes and E-cigarettes Among Dual Users
Brief Title: Nicotine Regulation for Dual Users of E-cigarettes and Cigarettes
Acronym: RDEC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Elias Klemperer, Assistant Professor, University of Vermont
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: R01DA059562 (NIH)
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2024-09

CONDITIONS: Tobacco Use Disorder
Keywords: Cigarettes; E-cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Vaping

STUDY DESIGN:
Intervention Model Description: 2x2 factorial randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- RC 1 + REC 1 (Experimental): Research cigarettes #1 plus research e-cigarettes #1
  Interventions: Other: Varying the nicotine content of cigarettes; Other: Varying the nicotine content of e-cigarettes
- RC 1 + REC 2 (Experimental): Research cigarettes #1 plus research e-cigarettes #2
  Interventions: Other: Varying the nicotine content of cigarettes; Other: Varying the nicotine content of e-cigarettes
- RC 2 + REC 1 (Experimental): Research cigarettes #2 plus research cigarettes #1
  Interventions: Other: Varying the nicotine content of cigarettes; Other: Varying the nicotine content of e-cigarettes
- RC 2 + REC 2 (Experimental): Research cigarettes #2 + research e-cigarettes #2
  Interventions: Other: Varying the nicotine content of cigarettes; Other: Varying the nicotine content of e-cigarettes

INTERVENTIONS:
Other: Varying the nicotine content of cigarettes — Altering the nicotine content of the tobacco research cigarettes
  Other Names: Comparing normal nicotine content (RC 1) to very low nicotine content (RC 2)
Other: Varying the nicotine content of e-cigarettes — Altering the nicotine content of the research e-cigarettes
  Other Names: Comparing high nicotine content (REC 1) to low nicotine content (REC 2)

SUMMARY:
Cigarette smoking remains the leading cause of preventable morbidity and mortality in the US. Use of multiple tobacco products is becoming increasingly prevalent, with dual use of e-cigarettes and cigarettes representing the most common combination. Though e-cigarettes are not without risk, completely switching from cigarettes to e-cigarettes likely reduces risk for tobacco-related harm. However, many established dual users maintain long-term smoking and the majority who use e-cigarettes non-daily are at an even greater risk for prolonged smoking than exclusive cigarette smokers. The Food and Drug Administration Center for Tobacco Products (FDA CTP) has announced plans to implement a nicotine-limiting product standard, capping the nicotine in cigarettes at a minimally or non-addictive level. Randomized controlled trials (RCTs) demonstrate that adults who exclusively smoke cigarettes respond to very low nicotine content (VLNC) cigarettes with reductions in smoking, demand, and dependence. However, nicotine reduction RCTs to date have excluded people who regularly use e-cigarettes and therefore it remains unclear how a nicotine-limiting standard for cigarettes would affect smoking among dual users. Given the potential substitutability of e-cigarettes for cigarettes, reducing the nicotine in cigarettes could promote a transition to exclusive e-cigarette use among dual users unable to completely quit nicotine, but only if sufficiently appealing e-cigarettes remain available. E-cigarettes containing 5% nicotine-salt solution are currently most popular in the US, but policy makers have proposed restricting e-cigarettes to ≤ 2% nicotine to curb youth e-cigarette use, and several states have already set limits to reduce nicotine in e-cigarettes. Prior laboratory studies indicate that higher vs lower nicotine e-cigarettes serve as better substitutes for cigarettes among adult dual users. As such, a restriction on e-cigarette nicotine concentration could undermine the potential for e-cigarettes to substitute for cigarettes and diminish the benefits of a nicotine-limiting standard for cigarettes among dual users. This study is a 12-week double-blind 2 cigarette level (Normal Nicotine vs Very Low Nicotine) x 2 e-cigarette level (High Nicotine vs Low Nicotine) between-subjects factorial trial to investigate how a nicotine-limiting standard for cigarettes affects adult dual users and whether these effects are impacted by constraints on e-cigarette nicotine concentration. Outcome measures include cigarettes per day, cigarette dependence, and toxicant exposure. The research is highly relevant to FDA CTP domains of Addiction and Behavior because it will test whether reducing the nicotine content of cigarettes reduces smoking and dependence, and whether these effects are moderated by the availability of high vs low nicotine e-cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* Regular use of tobacco
* 21 year of age or older
* Speak, comprehend and read English well enough to complete study procedures

Exclusion Criteria:

* Pregnant, trying to become pregnant, or nursing
* Under the age of 21
* Health conditions that could undermine ability to complete the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of cigarettes smoked per day | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elias Klemperer, PhD, Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - Brown University, Providence, Rhode Island
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available once we have published the results of the parent trials and manuscripts based on secondary analyses of those data, which we anticipate taking approximately three years.
Supporting Information: Study Protocol, SAP, ICF